CLINICAL TRIAL: NCT06567626
Title: Mixed Methods Co-design and Evaluation of a DECIsion Support Tool to Enable Shared DEcision Making With People Who Are Considering Revascularisation Options for Coronary Artery Disease
Brief Title: Decision Support Tool for Revascularisation Options in Coronary Artery Disease
Acronym: DECIDE-CAD
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 1000; IRAS 338504 (Other: Health Research Authority)
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Shared Decision Making; Percutaneous Coronary Intervention (PCI); Coronary Artery Bypass Grafting (CABG)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DST Co-Design (Work Package 1): * 40 people with lived experience of coronary revascularisation
  * 38 healthcare professionals
- DST Feasibility (Work Package 2): * 40 people awaiting coronary revascularisation
  * 8 healthcare professionals
  Interventions: Other: Decision Support Tool (DECIDE-CAD)

INTERVENTIONS:
Other: Decision Support Tool (DECIDE-CAD) — DECIDE-CAD is a decision support tool - designed using mixed methods through this study - which aims to enable shared decision making with people who are considering revascularisation options for coronary artery disease.
  Groups: DST Feasibility (Work Package 2)

SUMMARY:
Together with patients and healthcare professionals, we want to design a Decision Support Tool (DST) that will help people with coronary artery disease to understand and choose treatments that best reflect their preferences and values.

Coronary artery disease (CAD) is a leading cause of death. Blood vessels supplying oxygen to the heart muscle become narrowed by a gradual build-up of fatty material. This can result in heart attacks, heart failure, and sudden death. One way to treat the blockage is by inserting an inner sleeve called a "stent" into the blood vessel and clearing the blockage by forcing it into the artery wall. Another method involves diverting the blood supply around the blockage using a vessel harvested from another body site; this is called "bypass surgery". The best treatment, either stents or surgery, is different for everyone.

A Decision Support Tool (DST) will provide key information on the pros and cons of stents or surgery and how these match an individual's preferences and values. People are then empowered to make shared decisions about treatment with their doctors. Personalising treatment decisions in this way can reduce inequalities in care and improve shared decision making. Our proposed research will develop a DST in the form of a webpage with alternative print material for those at risk of digital poverty. The DST will be developed in multiple languages to improve accessibility.

There are two parts to the study: the first part will use the experience of patients, who have already had stent or surgery, and healthcare professionals to design and refine a DST prototype; this will be done through workshops, focus groups, and cognitive interviews. The second part will test whether it is possible to use the DST by people with CAD waiting for a procedure; this will be done through questionnaires and interviews. The result of this study can then subsequently inform an assessment of the refined DST on a national level, with the hopes of enabling more effective shared decision making.

ELIGIBILITY:
WP1. DST CO-DESIGN PATIENT PARTICIPANTS

Inclusion Criteria

Participants may enter the study if ALL of the following applies:

1. Any adult (≥ 18 years) with lived experience of coronary revascularisation
2. Willing and able to consent to study participation.
3. Able to understand written and spoken English for decisional needs workshop or focus groups (NB this criterion is not required for cognitive interviews or acceptability questionnaire)

Exclusion Criteria

Participants may not enter the study if they are unable to provide informed consent. Individuals who participate in focus groups are ineligible for subsequent participation in cognitive interviews and acceptability questionnaires.

WP1. DST CO-DESIGN HCP PARTICIPANTS

Inclusion Criteria

Participants may enter the study if ALL of the following applies:

1. Healthcare professional with a patient-facing clinical role which involves decision making regarding coronary revascularisation
2. Willing and able to consent to study participation.
3. Able to understand written and spoken English

Exclusion Criteria

Participants may not enter the study if they are unable to provide informed consent.

WP2. DST FEASIBILITY PATIENT PARTICIPANTS

Inclusion Criteria

Participants may enter the study if ALL of the following applies:

1. Adult (≥ 18 years) awaiting coronary revascularisation
2. Has received coronary angiography for definitive diagnosis.
3. Willing and able to consent to study participation.
4. Able to understand written and spoken English, Polish, Romanian, Urdu, Panjabi, or Gujarati

Exclusion Criteria

Participants may not enter the trial if ANY of the following apply:

1. Where clinical consensus strongly recommends one option of revascularisation over another
2. Unable to provide informed consent
3. Unable to speak one of the aforementioned 6 languages

WP2. DST FEASIBILITY HCP PARTICIPANTS

Inclusion Criteria

Participants may enter the study if ALL of the following applies:

1. Healthcare professional with a patient-facing clinical role which involves decision making regarding coronary revascularisation
2. Willing and able to consent to study participation.
3. Able to understand written and spoken English

Exclusion Criteria

Participants may not enter the study if they are unable to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Work Package 1:
  * 40 people with lived experience of coronary revascularisation
  * 38 healthcare professionals
  Work Package 2:
  * 40 people awaiting coronary revascularisation
  * 8 healthcare professionals
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of eligibility | 6 months
  Eligibility will be calculated as all patients eligible for study participation as a proportion of all patients who receive ACS treatment during the study period.
Rate of enrolment | 6 months
  Enrolment will be calculated as patients who provide informed consent and receive the DST as a proportion of all eligible patients.
Rate of attrition | 6 months
  Attrition will be calculated as patients who do not complete the study as a proportion of all patients enrolled.

SECONDARY OUTCOMES:
Decisional Conflict | 6 weeks
  Level of decisional conflict, measured using Decisional Conflict Scale before and after revascularisation procedure.
Acceptability | 6 weeks
  User acceptability of decision support tool, measured using researcher-generated questionnaire after revascularisation procedure.
Knowledge | 6 weeks
  User knowledge about revascularisation options, measured using researcher-regenerated questionnaire before and after revascularisation procedure.
Preference | 6 weeks
  User preference about revascularisation options, measured using Control Preference Scale and Patients Preferences Questionnaire for Angina treatment before and after revascularisation procedure.
Satisfaction with decision | 6 weeks
  User satisfaction with decision, measured using Satisfaction with Decision Scale after revascularisation procedure.
Decision Regret | 6 weeks
  Degree of decision regret about revascularisation treatment received, measured using Decision Regret Scale after revascularisation procedure
Treatment concordance | 6 weeks
  Concordance between user's preferred procedure and the treatment received, assessed after revascularisation procedure.
Level of shared decision making | 6 weeks
  Level of shared decision making experienced by the user, measured using Shared Decision Making Questionnaire (SDM-Q-9) after revascularisation procedure.
Health status | 6 weeks
  Health status measured using 20-item Short Form Survey before and after revascularisation procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University of Leicester, Leicester
  - University Hospitals of Leicester, Leicester

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised individual participant data can be made available on request for future studies with ethics approval.
Supporting Information: Study Protocol
Access Criteria: Requests must be from studies with appropriate ethics approval in place.